CLINICAL TRIAL: NCT01769196
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Assess the Efficacy and Safety of Simtuzumab (GS-6624) in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Study to Assess the Efficacy and Safety of Simtuzumab (GS-6624) in Adults With Idiopathic Pulmonary Fibrosis (IPF)
Acronym: RAINIER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Study was terminated due to lack of efficacy.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-322-0207; 2012-001571-36 (EudraCT Number)
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic; Pulmonary; Fibrosis; IPF
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Fibrosis | interventions — simtuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Simtuzumab (Experimental): Participants will receive simtuzumab for up to 254 weeks.
  Interventions: Drug: Simtuzumab
- Simtuzumab Placebo (Placebo Comparator): Participants will receive simtuzumab placebo for up to 254 weeks.
  Interventions: Drug: Simtuzumab placebo

INTERVENTIONS:
Drug: Simtuzumab — 125 mg/mL single-dose vials administered subcutaneously once a week
  Other Names: GS-6624
  Arms: Simtuzumab
Drug: Simtuzumab placebo — Simtuzumab placebo single-dose vials administered subcutaneously once a week
  Arms: Simtuzumab Placebo

SUMMARY:
The primary objectives of this study are to determine the effect of simtuzumab (GS-6624) on progression-free survival (PFS) as determined by either a categorical decline in forced vital capacity (FVC) or all-cause mortality, in all participants enrolled or in a subset of participants who are classified as lysyl oxidase-like-2 (LOXL2) high based on a prespecified level in serum at baseline.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects from 45 to 85 years of age
* Definite IPF within 3 years prior to screening
* Be able to walk at least 50 meters

Key Exclusion Criteria:

* Significant diseases other than IPF
* Obstructive lung disease
* Aortic aneurysm greater than or equal to 3.5 cm in diameter
* Treatment with immunosuppressive, cytotoxic, or antifibrotic drugs < 28 days prior to randomization are not permitted.

  * N-acetylcysteine is permitted provided the individual has been on a stable dose for > 4 weeks prior to screening
  * Concomitant use of pirfenidone or nintedanib must be in accordance with the approved prescribing instructions in the country where the site is located
* Individuals actively listed for lung transplant are excluded. However individuals at transplant centers with long waiting times (greater than 1 year) may be permitted to enter the study after discussion with Medical Monitor.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2016-02-23 (Actual); Study Completion 2016-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (175):
- United States (72):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Pulmonary Specialists, Ltd., Phoenix, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arizona Pulmonary Specialists, Ltd., Scottsdale, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - The University of Arizona, Tucson, Arizona
  - University of California San Diego, La Jolla, California
  - David Geffen School of Medicine at University of California, Los Angeles, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Sansum Clinic, Santa Barbara, California
  - Stanford University Medical Center, Stanford, California
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Bay Area Chest Physicians, Clearwater, Florida
  - University of Florida, Jacksonville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Tampa General Hospital, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Southeastern Lung Care, Decatur, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Loess Hills Clinical Research Center, Council Bluffs, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Tufts University School of Medicine, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - CardioPulmonary Associates, Chesterfield, Missouri
  - Saint Luke's Midwest Pulmonary Consultants, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Pulmonary and Allergy Associates, PA, Summit, New Jersey
  - Albany Medical College, Albany, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - North Shore University Hospital, New Hyde Park, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - The Oregon Clinic, PC, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Temple Lung Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Presbyterian - Montefiore, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Providence Everett Medical Center, Everett, Washington
  - University of Washington, Seattle, Washington
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (10):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Saint Vincents Hospital, Darlinghurst, New South Wales
  - Mater Adult Hospital, Brisbane, Queensland
  - Prince Charles Hospital, Chermside, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Belgium (3):
  - ULB Erasme, Anderlecht, Brussels Capital
  - Universitair Ziekenhuis Leuven, Leuven, Flemish Brabant
  - Cliniques Universitaires UCL de Mont-Godinne, Yvoir, Namur
- Canada (7):
  - Kelowna Respiratory and Allergy Clinic, Kelowna, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of British Columbia, Vancouver, British Columbia
  - Saint Joseph's Healthcare, Hamilton, Ontario
  - University Health Network, Toronto, Ontario
  - Centre Hospitalier de L'Université de Montréal Hôtel-Dieu, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec
- Czechia (7):
  - Fakultní nemocnice Brno, Brno, Jihormoravsky Kraj
  - Nemocnice Jihlava, Jihlava, Jihormoravsky Kraj
  - Krajská nemocnice Liberec a.s., Liberec, Severocesky Kraj
  - Masarykova nemocnice v Ústí nad Labem o.z., Ústí nad Labem, Severocesky Kraj
  - Fakultní Nemocnice Ostrava, Ostrava - Poruba, Severomoravsky Kraj
  - Fakultní nemocnice Plzen, Pilsen, Zapadocesky Kraj
  - Thomayerova nemocnice, Prague 4 - Krc
- France (13):
  - Hôpitaux Universitaires de Strasbourg, Strasbourg, Alsace
  - Centre Hospitalier Universitaire Grenoble Hopital Michalon, Grenoble, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire de Rennes, Hôpital Pontchaillou, Rennes, Brittany Region
  - Centre Hospitalier Régional et Universitaire - Hôpital Bretonneau, Tours, Centre-Val de Loire
  - Hôpital Albert Calmette, Lille, Hauts-de-France
  - Hôpital Arnaud de Villeneuve, Montpellier, Languedoc-roussillon
  - Hôpital Larrey, CHU de Toulouse, Service de Pneumologie, Toulouse, Midi-pyrenees
  - Centre Hospitalier Universitaire de Nice-Hôpital Pasteur, Nice, Poitou-charentes
  - Centre Hospitalier Universitaire Hôpital Nord, Marseille, Provence-Alpes-Côte d'Azur Region
  - Hôpital Louis Pradel, Bron, Rhone-aples
  - Centre Hospitalier Universitaire Hôpital Avicenne, Bobigny, Île-de-France Region
  - Hôpital Bichat-Claude Bernard, Paris, Île-de-France Region
  - HEGP, Paris, Île-de-France Region
- Germany (10):
  - Universität Freiburg, Klinikum, Abt für Pneumologie, Freiburg im Breisgau, Baden-Wurttemberg
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Ruhrlandklinik, Mannheim, Baden-Wurttemberg
  - Klinikum Großhadern der Ludwig-Maximilians-Universität München, München, Bavaria
  - Philipps-Universität und Universitätsklinikum Gießen und Marburg GmbH, Giessen, Hesse
  - Lungenfachklinik Immenhausen, Immenhausen, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Fachkrankenhaus Coswig, Coswig, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Helios Klinikum Emil von Behring, Lungenklinik Heckeshorn, Berlin
- Israel (6):
  - Soroka University Medical Center, Beersheba, Beersheba
  - Chaim Sheba Medical Center, Tel Litwinsky, Tel Aviv
  - Hadassah-Hebrew University Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petach Tikvah
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (9):
  - Ospedale "G.B.Morgagni - L. Pierantoni", Forlì, Forli-cesena
  - Azienda Ospedaliera San Gerardo di Monza, Monza, Monza E Brianza
  - Policlinico Universitario di Catania, Catania
  - San Giuseppe Hospital, Dept. of Internal Medicine, Milan
  - Azienda Ospedaliero-Universitaria Policlinico di Modena, Modena
  - Università degli studi Federico II di Napoli, Napoli
  - Istituto Mediterraneo Trapianti e Terapia Alta Specializzazione (ISMETT), Palermo
  - Fondazione PTV - Policlinico Tor Vergata, Roma
  - Azienda Ospedaliera Universitaria Senese Policlinico Le Scotte, Siena
- Poland (5):
  - 10 Wojskowy Szpital Kliniczny z Poliklinika SP ZOZ w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Instytut Gruzlicy i Chorób Pluc, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 3 w Zabrzu Slaskiego Uniwersytetu Medycznego w Katowicach, Zabrze, Silesian Voivodeship
  - Samodzielny Publiczny ZOZ, Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego, Lódz, Łódź Voivodeship
- South Korea (7):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Samsung Medical Center, Seoul, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (7):
  - Hospital Quirón Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Switzerland (3):
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Centre Hospitalier Universitaire Vaudois Lausanne (CHUV), Lausanne, Canton of Vaud
  - Universitätsspital Basel, Basel
- United Kingdom (16):
  - Birmingham Heartlands Hospital, Birmingham, England
  - Southmead Hospital, Bristol, England
  - Papworth Hospital, Cambridge, England
  - Castle Hill Hospital, Cottingham, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Saint James's University Hospital, Leeds, England
  - Glenfield Hospital, Leicester, England
  - Aintree University Hospitals NHS Foundation Trust, Liverpool, England
  - Royal Brompton Hospital, London, England
  - University Hospital of South Manchester NHS Foundation Trust, Manchester, England
  - Nottingham City Hospital, Nottingham, England
  - Churchill Hospital, Oxford, England
  - Northern General Hospital, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - Glasgow Royal Infirmary, Glasgow, Scotland

REFERENCES:
- [Background] Raghu G, Brown KK, Collard HR, Cottin V, Gibson KF, Kaner RJ, Lederer DJ, Martinez FJ, Noble PW, Song JW, Wells AU, Whelan TP, Wuyts W, Moreau E, Patterson SD, Smith V, Bayly S, Chien JW, Gong Q, Zhang JJ, O'Riordan TG. Efficacy of simtuzumab versus placebo in patients with idiopathic pulmonary fibrosis: a randomised, double-blind, controlled, phase 2 trial. Lancet Respir Med. 2017 Jan;5(1):22-32. doi: 10.1016/S2213-2600(16)30421-0. Epub 2016 Dec 7. PMID 27939076
- [Result] Humphries SM, O'Riordan TG, Zhang JJ, Bayly S, Sood R, Hayden A, Lynch DA; Relationship Baseline Fibrosis Score to Lung Function in A Clinical Trial Population with Idiopathic Pulmonary Fibrosis. ATS International Conference, 2016 May 13-18, San Francisco CA.
- [Result] Raghu G, Brown K, Collard H, Lederer D, Martinez F, Noble P, Song JW, Wells A, Whelan T, Moreau E, Patterson S, Bayly S, Chien J, Zhang J, O'Riordan T; Simtuzumab in Idiopathic Pulmonary Fibrosis: Results of a Randomized Clinical Trial. ERS Congress, 2016 September 3-7, London, UK.
- [Result] Raghu G, Brown KK, Collard HR, Lederer DJ, Martinez FJ, Noble PW, Song JW, Wells AU, Whalen TP, Lambert L, Chien JW, Zhang JJ, O'Riordan TG; Simtuzumab in Idiopathic Pulmonary Fibrosis (IPF): Baseline Demographic and Lung Function Data from a Clinical Trial. ATS International Conference, 2016 May 13-18, San Francisco CA.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, and Asia Pacific. The first participant was screened on 31 January 2013. The last study visit occurred on 23 February 2016.
Pre-assignment Details: 1250 participants were screened.
Groups:
- Simtuzumab: Simtuzumab 125 mg/mL administered subcutaneously once a week
- Simtuzumab Placebo: Simtuzumab placebo administered subcutaneously once a week
Period: Overall Study
Arm/Group | Simtuzumab | Simtuzumab Placebo
Started | 272 | 272
Completed | 0 | 0
Not Completed | 272 | 272
Not completed — Adverse Event | 24 | 20
Not completed — Death | 21 | 26
Not completed — Investigator Discretion | 7 | 3
Not completed — Lack of Efficacy | 3 | 2
Not completed — Progressive disease | 11 | 6
Not completed — Protocol defined criteria for withdrawal | 9 | 11
Not completed — Protocol Violation | 0 | 3
Not completed — Study terminated by sponsor | 160 | 161
Not completed — Participant never dosed with study drug | 1 | 0
Not completed — Withdrew consent | 36 | 40

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Analysis Set included all participants who were randomized into the study, and were analyzed according to treatment randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Simtuzumab | Simtuzumab Placebo | Total
Number analyzed (Participants) | 272 | 272 | 544
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (7.60) | 68.5 (7.07) | 68.1 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 47 | 92
  Male | 227 | 225 | 452
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 35 | 36 | 71
  Black | 3 | 3 | 6
  White | 231 | 229 | 460
  Other | 3 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 267 | 264 | 531
  Not Permitted | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 102 | 106 | 208
  Korea, Republic of | 34 | 35 | 69
  Spain | 11 | 13 | 24
  Canada | 10 | 14 | 24
  Czech Republic | 6 | 6 | 12
  Belgium | 10 | 4 | 14
  United Kingdom | 12 | 21 | 33
  Poland | 15 | 13 | 28
  Italy | 8 | 6 | 14
  Israel | 7 | 5 | 12
  Australia | 11 | 18 | 29
  France | 24 | 12 | 36
  Germany | 22 | 18 | 40
  Switzerland | 0 | 1 | 1
Forced vital capacity (FVC) Percent Predicted [Mean (Standard Deviation); unit: FVC % predicted] | 61.4 (12.17) | 62.3 (12.22) | 61.8 (12.19)
FVC % Predicted Category [Count of Participants; unit: Participants]
  Mild | 37 | 46 | 83
  Moderate | 152 | 150 | 302
  Severe | 83 | 76 | 159
Baseline Serum LOXL2 [Mean (Standard Deviation); unit: pg/mL] | 89.8 (70.06) | 86.7 (51.99) | 88.2 (61.48)

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival (PFS) was defined as the categorical decrease in forced vital capacity (FVC) % predicted (≥ 10% relative decrease in FVC and ≥ 5% absolute decrease in FVC from baseline) with confirmation at a consecutive visit at least 2 weeks later using the same criteria.
Time Frame: Up to 148 weeks
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Simtuzumab | Simtuzumab Placebo
Number analyzed (Participants) | 272 | 272
months | 12.6 [11.3 to 14.4] | 15.4 [12.6 to 19.1]
Statistical Analysis 1: Comparison: Simtuzumab vs Simtuzumab Placebo; Test type: Superiority — The null hypothesis was that there is no difference in PFS between simtuzumab and simtuzumab placebo. The alternative hypothesis was that there is a difference. These hypotheses were evaluated using stratified log-rank test, adjusted for screening post-bronchodilator FVC % predicted, sLOXL2 level categories and concomitant use of pirfenidone or nintedanib (P/N) at time of screening; p = 0.329, Log Rank; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.88 to 1.45] — Hazard ratio was estimated from Cox regression model adjusted for treatment and stratified for screening post-bronchodilator FVC % predicted, sLOXL2 level categories, and concomitant pirfenidone/nintedanib use at time of screening

2. Primary Outcome: PFS Among the Participants With sLOXL2 ≥ 50th Percentile
Time Frame: Up to 148 weeks
Population: Participants in the ITT Analysis Set with serum LOXL2 (sLOXL2) ≥ 50th percentile in peripheral blood were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Simtuzumab | Simtuzumab Placebo
Number analyzed (Participants) | 137 | 140
months | 11.7 [9.9 to 15.9] | 14.3 [10.4 to 19.1]
Statistical Analysis 1: Comparison: Simtuzumab vs Simtuzumab Placebo; Test type: Superiority — The null hypothesis was that there is no difference in PFS between simtuzumab and simtuzumab placebo in participants with sLOXL2 ≥ 50th percentile. The alternative hypothesis was that there is a difference. These hypotheses were evaluated using stratified log-rank test, adjusted for screening post-bronchodilator FVC % predicted and concomitant use of pirfenidone or nintedanib (P/N) at time of screening; p = 0.851, Log Rank; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.74 to 1.43] — Hazard ratio was estimated from Cox regression model adjusted for treatment and stratified for screening post-bronchodilator FVC % predicted and concomitant pirfenidone/nintedanib use at time of screening

3. Primary Outcome: PFS Among the Participants With sLOXL2 ≥ 75th Percentile
Time Frame: Up to 148 weeks
Population: Participants in the ITT Analysis Set with sLOXL2 ≥ 75th percentile in peripheral blood were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Simtuzumab | Simtuzumab Placebo
Number analyzed (Participants) | 68 | 71
months | 11.6 [9.0 to 15.0] | 16.9 [7.7 to 21.7]
Statistical Analysis 1: Comparison: Simtuzumab vs Simtuzumab Placebo; Test type: Superiority — The null hypothesis was that there is no difference in PFS between simtuzumab and simtuzumab placebo in participants with sLOXL2 ≥ 75th percentile. The alternative hypothesis was that there is a difference. These hypotheses were evaluated using stratified log-rank test, adjusted for screening post-bronchodilator FVC % predicted and concomitant use of pirfenidone or nintedanib (P/N) at time of screening; p = 0.475, Log Rank; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.72 to 2.00] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from randomization date to death that occurred prior to the last dose date plus 30 days.
Time Frame: Up to 151 weeks
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Simtuzumab | Simtuzumab Placebo
Number analyzed (Participants) | 272 | 272
months | NA [NA to NA] — NA = Not reached due to insufficient number of events | NA [NA to NA] — NA = Not reached due to insufficient number of events
Statistical Analysis 1: Comparison: Simtuzumab vs Simtuzumab Placebo; Test type: Other; p = 0.602, Log Rank; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.61 to 2.37] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Overall Survival Among the Participants With sLOXL2 ≥ 50th Percentile
Time Frame: Up to 151 weeks
Population: Participants in the ITT Analysis Set with sLOXL2 ≥ 50th percentile in peripheral blood were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Simtuzumab | Simtuzumab Placebo
Number analyzed (Participants) | 137 | 140
months | NA [NA to NA] — NA = Not reached due to insufficient number of events | NA [NA to NA] — NA = Not reached due to insufficient number of events
Statistical Analysis 1: Comparison: Simtuzumab vs Simtuzumab Placebo; Test type: Other — The difference in OS between the treatment groups was assessed using the stratified log-rank test, adjusted for screening post-bronchodilator FVC % predicted and concomitant use of pirfenidone or nintedanib (P/N) at time of screening; p = 0.988, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.43 to 2.28] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Overall Survival Among the Participants With sLOXL2 ≥ 75th Percentile
Time Frame: Up to 151 weeks
Population: Participants in the ITT Analysis Set with sLOXL2 ≥ 75th percentile in peripheral blood were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Simtuzumab | Simtuzumab Placebo
Number analyzed (Participants) | 68 | 71
months | NA [19.2 to NA] — NA = Not reached due to insufficient number of events | NA [NA to NA] — NA = Not reached due to insufficient number of events
Statistical Analysis 1: Comparison: Simtuzumab vs Simtuzumab Placebo; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.925, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.30 to 2.99] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Relative Change From Baseline in FVC % Predicted
Description: * FVC was defined as the volume of air (liters) that can forcibly be blown out after taking a full breath. FVC % predicted was defined as FVC % of the participant divided by the average FVC % in the population for any person of similar age, sex, and body composition.
  * Adjusted means were from mixed model repeated measures (MMRM) model with baseline FVC % predicted, sLOXL2 level, concomitant pirfenidone/nintedanib use (never vs. ever), treatment, visit, and treatment-by-visit interaction terms, including all data up to Week 130
  * The relative change was calculated as 100% * ( value at later time point minus value at baseline ) / value at baseline, with lower values indicating a decrease and higher values indicating an increase.
Time Frame: Weeks 54, 106, and 130
Population: Participants in the ITT Analysis Set with available data were analyzed. Any participant with available outcome data on baseline or post-baseline was included in the MMRM model, thus all 272 participants in each of the two treatment groups were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: Percent change in FVC % predicted
Arm/Group | Simtuzumab | Simtuzumab Placebo
Number analyzed (Participants) | 272 | 272
Percent change in FVC % predicted
  Week 54: number analyzed (Participants) | 124 | 117
  Week 54 | -9.20 (0.643) | -8.88 (0.658)
  Week 106: number analyzed (Participants) | 60 | 55
  Week 106 | -13.70 (0.883) | -12.16 (0.908)
  Week 130: number analyzed (Participants) | 10 | 12
  Week 130 | -18.09 (1.712) | -11.83 (1.600)

8. Secondary Outcome: Definite Acute Exacerbations of IPF Among Adjudicated Respiratory Hospitalizations
Time Frame: Up to 148 weeks
Population: Participants in the ITT Analysis Set with adjudicated respiratory hospitalizations were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Simtuzumab | Simtuzumab Placebo
Number analyzed (Participants) | 99 | 84
Participants | 5 | 5

9. Secondary Outcome: Number of Adjudicated Respiratory Hospitalizations (ARP) Among Total Hospitalizations
Time Frame: Up to 148 weeks
Population: Participants in ITT Analysis Set with total hospitalizations were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Simtuzumab | Simtuzumab Placebo
Number analyzed (Participants) | 181 | 154
Participants | 99 | 84

10. Secondary Outcome: Number of Participants Experiencing Adjudicated Respiratory Deaths Among Those With Adjudicated Death
Time Frame: Up to 148 weeks
Population: Participants in the ITT Analysis Set with adjudicated deaths were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Simtuzumab | Simtuzumab Placebo
Number analyzed (Participants) | 19 | 17
Participants | 17 | 13

11. Secondary Outcome: Absolute Change From Baseline in 6 Minute Walk Distance (6MWD)
Description: * Adjusted means were from MMRM model with baseline 6MWD, FVC % predicted, sLOXL2 level, concomitant pirfenidone/nintedanib use (never vs. ever), treatment, visit, and treatment-by-visit interaction terms, including all data up to Week 130.
  * The absolute change was calculated as value at later time point minus value at baseline, with lower values indicating a decrease and higher values indicating an increase.
Time Frame: Weeks 58, 106, and 130
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Simtuzumab | Simtuzumab Placebo
Number analyzed (Participants) | 272 | 272
Meters
  Week 58: number analyzed (Participants) | 95 | 98
  Week 58 | -33.76 (6.617) | -14.70 (6.596)
  Week 106: number analyzed (Participants) | 44 | 37
  Week 106 | -37.43 (9.710) | -24.30 (10.318)
  Week 130: number analyzed (Participants) | 7 | 9
  Week 130 | -71.20 (19.140) | -31.65 (18.458)

12. Secondary Outcome: Absolute Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) Score
Description: * The SGRQ is a disease-specific questionnaire designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Patients respond to questions about symptoms (frequency & severity) and impact components (social functioning and psychological disturbances resulting from airways disease). Scores range from 0 to 100, with higher scores indicating more limitations.
  * The absolute change was calculated as value at later time point minus value at baseline, with lower values indicating a decrease and higher values indicating an increase.
Time Frame: Week 58, 106, and 130
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Simtuzumab | Simtuzumab Placebo
Number analyzed (Participants) | 272 | 272
units on a scale
  Week 58: number analyzed (Participants) | 101 | 104
  Week 58 | 6.07 (1.015) | 3.62 (1.010)
  Week 106: number analyzed (Participants) | 48 | 37
  Week 106 | 10.34 (1.425) | 6.54 (1.559)
  Week 130: number analyzed (Participants) | 10 | 10
  Week 130 | 18.10 (2.424) | 1.08 (2.473)

ADVERSE EVENTS:
Time Frame: 30 days post last study treatment (up to 148 weeks)
Description: Safety Analysis Set included all randomized participants who received at least 1 dose of study drug and was analyzed according to treatment received.
Arm/Group | Simtuzumab | Simtuzumab Placebo
All-Cause Mortality (participants affected / at risk) | 31/271 | 32/272
Serious Adverse Events (participants affected / at risk) | 101/271 | 97/272
Other Adverse Events (participants affected / at risk) | 237/271 | 246/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simtuzumab (N=271) | Simtuzumab Placebo (N=272)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 3 | 5
Acute right ventricular failure (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 2 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 6 | 1
Atrial flutter (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 3
Coronary artery occlusion (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pleuropericarditis (Cardiac disorders) | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Mesenteric venous occlusion (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 2
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 3
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 4 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Hepatic mass (Hepatobiliary disorders) | 0 | 1
Hepatic necrosis (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Hepatitis E (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 4
Lung infection (Infections and infestations) | 0 | 1
Mycetoma mycotic (Infections and infestations) | 0 | 1
Oropharyngitis fungal (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 16 | 18
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory moniliasis (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 3
Sepsis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Urosepsis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Post procedural stroke (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 2
VIth nerve paralysis (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 1 | 0
Goodpasture's syndrome (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 31 | 35
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 2 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Femoral artery occlusion (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simtuzumab (N=271) | Simtuzumab Placebo (N=272)
Constipation (Gastrointestinal disorders) | 16 | 13
Diarrhoea (Gastrointestinal disorders) | 44 | 47
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 21 | 22
Nausea (Gastrointestinal disorders) | 33 | 35
Asthenia (General disorders) | 15 | 17
Chest pain (General disorders) | 18 | 16
Fatigue (General disorders) | 49 | 48
Injection site bruising (General disorders) | 17 | 10
Oedema peripheral (General disorders) | 21 | 12
Pyrexia (General disorders) | 21 | 12
Bronchitis (Infections and infestations) | 32 | 39
Lower respiratory tract infection (Infections and infestations) | 8 | 15
Nasopharyngitis (Infections and infestations) | 36 | 43
Respiratory tract infection (Infections and infestations) | 14 | 17
Sinusitis (Infections and infestations) | 16 | 14
Upper respiratory tract infection (Infections and infestations) | 57 | 57
Weight decreased (Investigations) | 25 | 24
Decreased appetite (Metabolism and nutrition disorders) | 29 | 34
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 28
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 14
Dizziness (Nervous system disorders) | 31 | 26
Headache (Nervous system disorders) | 32 | 35
Depression (Psychiatric disorders) | 14 | 12
Insomnia (Psychiatric disorders) | 15 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 102 | 93
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 98 | 73
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 30 | 29
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 9
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 33 | 27
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 15
Productive cough (Respiratory, thoracic and mediastinal disorders) | 22 | 18
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 19 | 15
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 14 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 8
Rash (Skin and subcutaneous tissue disorders) | 22 | 21
Hypertension (Vascular disorders) | 15 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years